CLINICAL TRIAL: NCT07154043
Title: Comparison of Intermittent Pneumatic Compression Therapy as an Alternative or an Adjunct to Manual Lymphatic Drainage Within Complete Decongestive Therapy for Breast Cancer-Related Lymphedema
Brief Title: Comparison of IPC Therapy as an Alternative or an Adjunct to MLD Within CDT for BCRL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Oya Topuz, Professor Doctor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PamukkaleU.ftr-OTopuz-001
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer-Related Lymphedema; BCRL
Keywords: Breast Cancer-Related Lymphedema; Manual Lymph Drainage; Intermittent Pneumatic Compression; Complete Decongestive Therapy
MeSH Terms: conditions — Breast Cancer Lymphedema | interventions — carbohydrate-deficient transferrin; Manual Lymphatic Drainage

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Complete Decongestive Therapy plus Intermittent Pneumatic Compression Group (Experimental): Complete decongestive therapy program consisting of manual lymph drainage, multilayer bandaging, skin care, and exercise. In addition, patients will receive intermittent pneumatic compression with a device at 20-50 mmHg pressure for 40 minutes per session. The total treatment duration will be 115 minutes per session, 5 sessions per week, for 3 weeks.
  Interventions: Procedure: CDT + Intermittent Pneumatic Compression (IPC)
- Complete Decongestive Therapy without Manual Lymph Drainage plus Intermittent Pneumatic Compression (Experimental): This group will receive a complete decongestive therapy program consisting of multilayer bandaging, skin care, and exercise. Manual lymph drainage will be replaced by intermittent pneumatic compression. Intermittent pneumatic compression will be applied with a device at 20-50 mmHg pressure for 40 minutes per session. The total treatment duration will be 75 minutes per session, 5 sessions per week, for 3 weeks.
  Interventions: Procedure: CDT without Manual Lymph Drainage plus Intermittent Pneumatic Compression
- Complete Decongestive Therapy Group (Active Comparator): This group will receive a complete decongestive therapy program consisting of manual lymph drainage, multilayer bandaging, skin care, and exercise. The treatment duration will be 75 minutes per session, 5 sessions per week, for 3 weeks.
  Interventions: Procedure: Complete Decongestive Therapy (CDT)

INTERVENTIONS:
Procedure: Complete Decongestive Therapy (CDT) — Manual lymph drainage, multilayer bandaging, skin care, and exercise. 75 minutes per session, 5 sessions per week, for 3 weeks.
  Arms: Complete Decongestive Therapy Group
Procedure: CDT + Intermittent Pneumatic Compression (IPC) — Complete decongestive therapy program including manual lymph drainage, multilayer bandaging, skin care, and exercise, plus intermittent pneumatic compression at 20-50 mmHg for 40 minutes per session. Total duration: 115 minutes per session, 5 sessions per week, for 3 weeks.
  Arms: Complete Decongestive Therapy plus Intermittent Pneumatic Compression Group
Procedure: CDT without Manual Lymph Drainage plus Intermittent Pneumatic Compression — Complete decongestive therapy consisting of multilayer bandaging, skin care, and exercise, with manual lymph drainage replaced by intermittent pneumatic compression at 20-50 mmHg for 40 minutes per session. Total duration: 75 minutes per session, 5 sessions per week, for 3 weeks.
  Arms: Complete Decongestive Therapy without Manual Lymph Drainage plus Intermittent Pneumatic Compression

SUMMARY:
Breast cancer is the most common cancer among women worldwide and lymphedema is one of its most significant complications. Breast cancer-related lymphedema (BCRL) may develop shortly after treatment or even years later, causing physical and psychological burden, functional impairment, and reduced quality of life. Complete decongestive therapy (CDT), which includes manual lymph drainage (MLD), compression, skin care, and exercise, is the standard approach. Intermittent pneumatic compression (IPC) has been proposed as an additional option, and current consensus reports emphasize the need for studies evaluating IPC in combination with MLD.

Previous studies comparing IPC and MLD, either alone or in combination, have shown inconsistent results. Some reported no significant difference between treatment groups, while others suggested additional benefits of IPC, particularly in reducing limb heaviness and tension. However, there is still insufficient evidence to clarify the exact role of IPC within CDT.

The aim of this study is to investigate the acute effects of using IPC instead of MLD, or in combination with MLD, on arm circumference, arm volume, shoulder range of motion, and quality of life in patients with BCRL.

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy among women worldwide and remains the leading cause of cancer-related mortality in women. Breast cancer-related lymphedema (BCRL) is one of the most important complications of breast cancer treatment. It may occur due to lymphatic system damage caused by surgery and/or radiotherapy, or as a result of tumor-related lymphangiogenesis, leading to interstitial fluid accumulation. BCRL can develop immediately after treatment or months to years later.

BCRL is associated with swelling, heaviness, discomfort, weakness, increased risk of infection, and progressive chronicity, which together result in upper extremity dysfunction and reduced quality of life. Compared with women without lymphedema, patients with BCRL report more frequent pain, decreased shoulder mobility, reduced upper extremity strength, impaired daily activities, and sensory disturbances.

The standard treatment for BCRL is complete decongestive therapy (CDT), which consists of manual lymph drainage (MLD), compression, skin care, and exercise. Intermittent pneumatic compression (IPC) has also been proposed as a treatment option, and the 2023 consensus report of the International Society of Lymphology emphasized the need for further studies evaluating IPC in combination with MLD.

However, the number of studies directly comparing IPC with MLD, or evaluating their combined use, is limited and results remain inconsistent. Some trials reported no significant difference between MLD and IPC in terms of limb volume reduction, while others demonstrated additional benefits of IPC in relieving heaviness and tension. The role of IPC in CDT, whether as a replacement for MLD or as an adjunct, is not yet clearly defined.

The purpose of this study is to investigate the acute effects of using IPC instead of MLD, or in combination with MLD, within CDT on arm circumference, arm volume, shoulder range of motion, and quality of life in patients with BCRL.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Patients aged 18-65 years
* Having a history of unilateral mastectomy and lymph node dissection at least one year ago due to breast cancer diagnosis.
* Having unilateral breast cancer-related upper extremity lymphedema (>20% volume difference between the two upper extremities or >2 cm difference in circumference at any measured point) according to the diagnostic criteria of the International Society of Lymphology (Committee 2023) for at least six months.
* Not having received lymphedema treatment or exercise therapy for the last six months
* Completing breast cancer primary treatment at least 6 months ago (except hormone therapy/aromatase inhibitors)

Exclusion Criteria:

* Bilateral breast cancer
* Bilateral axillary lymph node dissection
* Metastatic breast cancer
* Receiving ongoing radiotherapy or chemotherapy
* Primary or bilateral lymphedema
* Having active cancer
* Presence of stage 3 lymphedema
* Uncontrolled serious systemic disease (cardiopulmonary diseases, arterial or venous diseases, renal dysfunction, uncontrolled hypertension or hypotension, cardiac arrhythmia, scleroderma, Sudek's atrophy).
* Current or recent (within the last 3 months) infection (cellulitis, lymphangitis) or deep venous thrombosis
* Presence of open wounds
* Using medications that may affect body fluid and electrolyte balance (diuretics, etc.).
* Individuals with serious mental and sensory problems
* Being pregnant
* Body mass index >40 kg/m2

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Arm volumetric measurements | 1 day before rehabilitation and 3 weeks after the start of rehabilitation
  Arm volume will be calculated using circumferential measurements taken with a standard 7 mm measuring tape at 4 cm intervals along the arm. Segmental arm volumes (mL-cm³) will be calculated using the simplified frustum formula (Frustum Model). This formula, as described by Sitzia et al., has shown high correlation with water displacement measurements and is widely used in the literature as a valid and reliable indirect method for assessing lymphedema.

SECONDARY OUTCOMES:
Shoulder Range of Motion | 1 day before rehabilitation and 3 weeks after the start of rehabilitation
  Goniometric measurements of the affected shoulder will be performed to assess flexion, extension, abduction, adduction, internal rotation, and external rotation in patients with lymphedema.
Quality of Life Measurement ULL-27 | 1 day before rehabilitation and 3 weeks after the start of rehabilitation
  ULL-27 quality of life questionnaire, developed specifically for upper extremity lymphedema patients. The scale has physical, psychological and social dimensions. It consists of 27 questions. A high score on the scale indicates that lymphedema negatively affects the quality of life.
Arm Circumference Measurements | 1 day before rehabilitation and 3 weeks after the start of rehabilitation
  To assess lymphedema severity, circumferential measurements of the affected and unaffected upper extremities will be performed. Patients' forearms will be in a supine position, elbows fully extended, and arms abducted at 90 degrees. Arm-hand circumference will be measured at four points: metacarpal region, wrist, 10 cm below the lateral epicondyle, and 15 cm above the lateral epicondyle, using a non-stretchable 7 mm tape of 150 cm length. Measurements will be taken on both upper extremities, and the differences between sides will be recorded in centimeters.
Quick Disabilities of the Arm, Shoulder, and Hand (Quick-DASH) Questionnaire | 1 day before rehabilitation and 3 weeks after the start of rehabilitation
  The Quick-DASH is an 11-item questionnaire used to assess activity limitations of the upper extremity in patients with lymphedema related to breast cancer. Each item is scored from 1 to 5, and total scores are summed. A total score of 0 indicates no disability, while a score of 100 indicates the highest level of disability. The Turkish version was validated in 2011 and has been found valid and reliable for assessing upper extremity activity limitations in breast cancer-related lymphedema.
Upper Extremity Swelling (Visual Analog Scale) | 1 day before rehabilitation and 3 weeks after the start of rehabilitation
  Swelling in the affected extremity will be assessed using a 0-10 cm (0-100 mm) horizontal Visual Analog Scale (VAS). A score of 0 indicates no symptom, and 10 cm indicates the most severe presence of the symptom. Participants will mark the severity of each symptom and the discomfort caused by the symptom on the VAS ("0" = no complaint, "10" = maximal complaint). The mark will be measured in centimeters with a ruler. The VAS is a valid and reliable method for measuring experimental and clinical pain as well as lymphedema-specific symptoms, and it is sensitive to small changes in symptom intensity.
Upper Extremity Heaviness (Visual Analog Scale) | 1 day before rehabilitation and 3 weeks after the start of rehabilitation
  Heaviness in the affected extremity will be assessed using a 0-10 cm (0-100 mm) horizontal Visual Analog Scale (VAS). A score of 0 indicates no symptom, and 10 cm indicates the most severe presence of the symptom. Participants will mark the severity of each symptom and the discomfort caused by the symptom on the VAS ("0" = no complaint, "10" = maximal complaint). The mark will be measured in centimeters with a ruler. The VAS is a valid and reliable method for measuring experimental and clinical pain as well as lymphedema-specific symptoms, and it is sensitive to small changes in symptom intensity.
Upper Extremity Tightness (Visual Analog Scale) | 1 day before rehabilitation and 3 weeks after the start of rehabilitation
  Tightness in the affected extremity will be assessed using a 0-10 cm (0-100 mm) horizontal Visual Analog Scale (VAS). A score of 0 indicates no symptom, and 10 cm indicates the most severe presence of the symptom. Participants will mark the severity of each symptom and the discomfort caused by the symptom on the VAS ("0" = no complaint, "10" = maximal complaint). The mark will be measured in centimeters with a ruler. The VAS is a valid and reliable method for measuring experimental and clinical pain as well as lymphedema-specific symptoms, and it is sensitive to small changes in symptom intensity.
Upper Extremity Pain (Visual Analog Scale) | 1 day before rehabilitation and 3 weeks after the start of rehabilitation
  Pain in the affected extremity will be assessed using a 0-10 cm (0-100 mm) horizontal Visual Analog Scale (VAS). A score of 0 indicates no symptom, and 10 cm indicates the most severe presence of the symptom. Participants will mark the severity of each symptom and the discomfort caused by the symptom on the VAS ("0" = no complaint, "10" = maximal complaint). The mark will be measured in centimeters with a ruler. The VAS is a valid and reliable method for measuring experimental and clinical pain as well as lymphedema-specific symptoms, and it is sensitive to small changes in symptom intensity.
Patient Satisfaction | 3 weeks after the start of rehabilitation
  Patient satisfaction with the exercise programs will be assessed using a 4-point Likert scale (0 = not satisfied, 1 = slightly satisfied, 2 = satisfied, 3 = very satisfied).
Perceived Improvement | 3 weeks after the start of rehabilitation
  Patients' perceived improvement will be measured using the Patient Global Perceived Improvement Scale, asking participants to compare their current condition with baseline regarding lymphedema (1 = much better, 2 = better, 3 = slightly better, 4 = no change, 5 = slightly worse, 6 = worse, 7 = much worse). The Turkish version of this scale was validated and culturally adapted by Yalçın et al. in 2003, showing good internal consistency (Cronbach's α = 0.79) and test-retest reliability (ICC = 0.75).

CONTACTS AND LOCATIONS:
Overall Officials: Oya Topuz, Professor, Study Director — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gummesson C, Ward MM, Atroshi I. The shortened disabilities of the arm, shoulder and hand questionnaire (QuickDASH): validity and reliability based on responses within the full-length DASH. BMC Musculoskelet Disord. 2006 May 18;7:44. doi: 10.1186/1471-2474-7-44. PMID 16709254
- [Background] LeBlanc M, Stineman M, DeMichele A, Stricker C, Mao JJ. Validation of QuickDASH outcome measure in breast cancer survivors for upper extremity disability. Arch Phys Med Rehabil. 2014 Mar;95(3):493-8. doi: 10.1016/j.apmr.2013.09.016. Epub 2013 Oct 2. PMID 24095658
- [Background] Koldas Dogan S, Ay S, Evcik D, Baser O. Adaptation of Turkish version of the questionnaire Quick Disability of the Arm, Shoulder, and Hand (Quick DASH) in patients with carpal tunnel syndrome. Clin Rheumatol. 2011 Feb;30(2):185-91. doi: 10.1007/s10067-010-1470-y. Epub 2010 Apr 22. PMID 20411289
- [Background] Sitzia J. Volume measurement in lymphoedema treatment: examination of formulae. Eur J Cancer Care (Engl). 1995 Mar;4(1):11-6. doi: 10.1111/j.1365-2354.1995.tb00047.x. PMID 7620649
- [Background] Karges JR, Mark BE, Stikeleather SJ, Worrell TW. Concurrent validity of upper-extremity volume estimates: comparison of calculated volume derived from girth measurements and water displacement volume. Phys Ther. 2003 Feb;83(2):134-45. PMID 12564949
- [Background] Executive Committee of the International Society of Lymphology. The diagnosis and treatment of peripheral lymphedema: 2020 Consensus Document of the International Society of Lymphology. Lymphology. 2020;53(1):3-19. PMID 32521126
- [Background] De Vrieze T, Gebruers N, Tjalma WA, Nevelsteen I, Thomis S, De Groef A, Dams L, Van der Gucht E, Belgrado JP, Vandermeeren L, Devoogdt N. What is the best method to determine excessive arm volume in patients with breast cancer-related lymphoedema in clinical practice? Reliability, time efficiency and clinical feasibility of five different methods. Clin Rehabil. 2019 Jul;33(7):1221-1232. doi: 10.1177/0269215519835907. Epub 2019 Mar 18. PMID 30880473
- [Background] Keeley V, Riches K, Ward L, Franks PJ. A Prospective Preliminary Study Examining the Physiological Impact of Pneumatic Compression Dosing in the Treatment of Lower Extremity Lymphedema. Lymphat Res Biol. 2023 Oct;21(5):456-462. doi: 10.1089/lrb.2022.0087. Epub 2023 May 4. PMID 37140559
- [Background] Kayali Vatansever A, Yavuzsen T, Karadibak D. The Reliability and Validity of Quality of Life Questionnaire Upper Limb Lymphedema (ULL-27) Turkish Patient With Breast Cancer Related Lymphedema. Front Oncol. 2020 May 12;10:455. doi: 10.3389/fonc.2020.00455. eCollection 2020. PMID 32477925
- [Background] Yalcin I, Bump RC. Validation of two global impression questionnaires for incontinence. Am J Obstet Gynecol. 2003 Jul;189(1):98-101. doi: 10.1067/mob.2003.379. PMID 12861145
- [Background] Stanton AW, Badger C, Sitzia J. Non-invasive assessment of the lymphedematous limb. Lymphology. 2000 Sep;33(3):122-35. PMID 11019400
- [Background] Szuba A, Achalu R, Rockson SG. Decongestive lymphatic therapy for patients with breast carcinoma-associated lymphedema. A randomized, prospective study of a role for adjunctive intermittent pneumatic compression. Cancer. 2002 Dec 1;95(11):2260-7. doi: 10.1002/cncr.10976. PMID 12436430
- [Background] Szolnoky G, Lakatos B, Keskeny T, Varga E, Varga M, Dobozy A, Kemeny L. Intermittent pneumatic compression acts synergistically with manual lymphatic drainage in complex decongestive physiotherapy for breast cancer treatment-related lymphedema. Lymphology. 2009 Dec;42(4):188-94. PMID 20218087
- [Background] Tastaban E, Soyder A, Aydin E, Sendur OF, Turan Y, Ture M, Bilgen M. Role of intermittent pneumatic compression in the treatment of breast cancer-related lymphoedema: a randomized controlled trial. Clin Rehabil. 2020 Feb;34(2):220-228. doi: 10.1177/0269215519888792. Epub 2019 Dec 4. PMID 31795748
- [Background] Uzkeser H, Karatay S, Erdemci B, Koc M, Senel K. Efficacy of manual lymphatic drainage and intermittent pneumatic compression pump use in the treatment of lymphedema after mastectomy: a randomized controlled trial. Breast Cancer. 2015 May;22(3):300-7. doi: 10.1007/s12282-013-0481-3. Epub 2013 Aug 8. PMID 23925581
- [Background] Sanal-Toprak C, Ozsoy-Unubol T, Bahar-Ozdemir Y, Akyuz G. The efficacy of intermittent pneumatic compression as a substitute for manual lymphatic drainage in complete decongestive therapy in the treatment of breast cancer related lymphedema. Lymphology. 2019;52(2):82-91. PMID 31525829
- [Background] Ridner SH, Fu MR, Wanchai A, Stewart BR, Armer JM, Cormier JN. Self-management of lymphedema: a systematic review of the literature from 2004 to 2011. Nurs Res. 2012 Jul-Aug;61(4):291-9. doi: 10.1097/NNR.0b013e31824f82b2. PMID 22565103
- [Background] Executive Committee of the International Society of Lymphology. The Diagnosis and Treatment of Peripheral Lymphedema: 2023 Consensus Document of The International Society of Lymphology. Lymphology. 2023;56(4):133-151. PMID 39207406
- [Background] Gursen C, Dylke ES, Moloney N, Meeus M, De Vrieze T, Devoogdt N, De Groef A. Self-reported signs and symptoms of secondary upper limb lymphoedema related to breast cancer treatment: Systematic review. Eur J Cancer Care (Engl). 2021 Sep;30(5):e13440. doi: 10.1111/ecc.13440. Epub 2021 Mar 18. PMID 33733550
- [Background] Orhan C, Uzelpasaci E, Baran E, Nakip G, Ozgul S, Aksoy S, Akbayrak T. The Reliability and Validity of the Turkish Version of the Lymphedema Life Impact Scale in Patients With Breast Cancer-Related Lymphedema. Cancer Nurs. 2020 Sep/Oct;43(5):375-383. doi: 10.1097/NCC.0000000000000709. PMID 30921030
- [Background] Smoot B, Wong J, Cooper B, Wanek L, Topp K, Byl N, Dodd M. Upper extremity impairments in women with or without lymphedema following breast cancer treatment. J Cancer Surviv. 2010 Jun;4(2):167-78. doi: 10.1007/s11764-010-0118-x. Epub 2010 Apr 7. PMID 20373044
- [Background] Lee TS, Morris CM, Czerniec SA, Mangion AJ. Does Lymphedema Severity Affect Quality of Life? Simple Question. Challenging Answers. Lymphat Res Biol. 2018 Feb;16(1):85-91. doi: 10.1089/lrb.2016.0049. Epub 2017 Apr 28. PMID 28453410
- [Background] Pinto M, Gimigliano F, Tatangelo F, Megna M, Izzo F, Gimigliano R, Iolascon G. Upper limb function and quality of life in breast cancer related lymphedema: a cross-sectional study. Eur J Phys Rehabil Med. 2013 Oct;49(5):665-73. Epub 2013 May 23. PMID 23698473
- [Background] Park JE, Jang HJ, Seo KS. Quality of life, upper extremity function and the effect of lymphedema treatment in breast cancer related lymphedema patients. Ann Rehabil Med. 2012 Apr;36(2):240-7. doi: 10.5535/arm.2012.36.2.240. Epub 2012 Apr 30. PMID 22639749
- [Background] Dawes DJ, Meterissian S, Goldberg M, Mayo NE. Impact of lymphoedema on arm function and health-related quality of life in women following breast cancer surgery. J Rehabil Med. 2008 Aug;40(8):651-8. doi: 10.2340/16501977-0232. PMID 19020699
- [Background] DiSipio T, Rye S, Newman B, Hayes S. Incidence of unilateral arm lymphoedema after breast cancer: a systematic review and meta-analysis. Lancet Oncol. 2013 May;14(6):500-15. doi: 10.1016/S1470-2045(13)70076-7. Epub 2013 Mar 27. PMID 23540561
- [Background] Pappalardo M, Starnoni M, Franceschini G, Baccarani A, De Santis G. Breast Cancer-Related Lymphedema: Recent Updates on Diagnosis, Severity and Available Treatments. J Pers Med. 2021 May 12;11(5):402. doi: 10.3390/jpm11050402. PMID 34065795
- [Background] McDuff SGR, Mina AI, Brunelle CL, Salama L, Warren LEG, Abouegylah M, Swaroop M, Skolny MN, Asdourian M, Gillespie T, Daniell K, Sayegh HE, Naoum GE, Zheng H, Taghian AG. Timing of Lymphedema After Treatment for Breast Cancer: When Are Patients Most At Risk? Int J Radiat Oncol Biol Phys. 2019 Jan 1;103(1):62-70. doi: 10.1016/j.ijrobp.2018.08.036. Epub 2018 Aug 28. PMID 30165125
- [Background] Mortimer P. Arm lymphoedema after breast cancer. Lancet Oncol. 2013 May;14(6):442-3. doi: 10.1016/S1470-2045(13)70097-4. Epub 2013 Mar 27. No abstract available. PMID 23540560
- [Background] Burckhardt M, Belzner M, Berg A, Fleischer S. Living with breast cancer-related lymphedema: a synthesis of qualitative research. Oncol Nurs Forum. 2014 Jul 1;41(4):E220-37. doi: 10.1188/14.ONF.E220-E237. PMID 24969257